CLINICAL TRIAL: NCT05875636
Title: GLP-1 Receptor Agonist Use and Incidence of Retained Gastric Food on Endoscopy
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Phillip Wilson, Principal Investigator/ Assistant Professor, Medical University of South Carolina
Other Study IDs: Pro00129059
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gastric Content Aspiration
MeSH Terms: conditions — Respiratory Aspiration of Gastric Contents | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients taking a GLP-1 agonist medication: Participants meeting all inclusion/exclusion criteria who are taking a GLP-1 agonist medication
  Interventions: Other: Esophagogastroduodenoscopy
- Controls: Participants meeting all inclusion/exclusion criteria and are NOT taking a GLP-1 agonist medication.
  Interventions: Other: Esophagogastroduodenoscopy

INTERVENTIONS:
Other: Esophagogastroduodenoscopy — All patients will undergo an esophagogastroduodenoscopy per standard of care, as scheduled.

SUMMARY:
This study will enroll patients ages 18 and over who are in one of the following groups 1) taking a GLP-1 receptor agonist medication 2) not taking a GLP-1 receptor agonist (control group), are undergoing EGS and have appropriately fasted. Study data will be collected in the form of qualitatively observing whether the stomach is empty as expected, or contains solid or clinically relevant liquid contents.

ELIGIBILITY:
Inclusion Criteria

* Adults 18 years of age and older presenting for esophagogastroduodenoscopy (EGD)
* One of the following groups:

  * GLP-1 receptor agonist cohort: active treatment with any GLP-1 receptor agonist therapy within prior 30 days
  * Control cohort: not taking a GLP-1 receptor agonist medication
* Appropriately fasted per ASA Fasting Guidelines

Exclusion Criteria

* Simultaneous bowel preparation/planned dual endoscopy with colonoscopy
* Any pre-planned alteration to standard fasting guidelines (ASA NPO guidelines)
* Emergency endoscopic procedure
* Concern for active GI bleeding
* Food impaction/foreign body as indication for procedure
* Gastric outlet obstruction/bowel obstruction
* Achalasia
* Zenker's diverticulum
* History of esophageal or gastric surgery
* Active pregnancy
* Chronic daily opioid therapy ≥ 15 MMEs per day
* Prokinetic agent use (i.e. metoclopramide)
* Inability or unwillingness of subject to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of patients who have appropriately fasted, and are scheduled for an esophagogastroduodenoscopy (EGD). Patients will fall in to two groups: 1) taking a GLP-1 receptor agonist or 2) not taking a receptor agonist medication.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Retained gastric food | From time of enrollment until the end of surgery, assessed up to 4 weeks
  Incidence of clinically significant retained gastric food, defined as visible solid/particulate matter, or liquid volume > 1.5cc/kg

SECONDARY OUTCOMES:
Incidence of pulmonary aspiration event | From the time surgery begins until the end of scheduled surgery, assessed up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Phillip R Wilson, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States